CLINICAL TRIAL: NCT03506789
Title: Dexamethasone Twice for Pain Treatment of Total Knee Arthroplasty - A Randomized Blinded Placebo-controlled Clinical Trial
Brief Title: Dexamethasone Twice for Pain Treatment of Total Knee Arthroplasty
Acronym: DEX-2-TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-KAKG-2018
Record Dates: First submitted 2018-02-21; First posted 2018-04-24 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A: (Active Comparator): 24 mg dexamethasone i.v. perioperatively and 24 mg dexamethasone i.v. on the first postoperative day
  Interventions: Drug: Dexamethasone
- Treatment B: (Active Comparator): 24 mg dexamethasone i.v. perioperatively and placebo (isotonic saline) i.v. on the first postoperative day
  Interventions: Drug: Dexamethasone; Drug: Placebos
- Placebo (Placebo Comparator): Placebo (isotonic saline) i.v. perioperatively and placebo (isotonic saline) i.v. on the first postoperative day
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 24 mg
  Arms: Treatment A:; Treatment B:
Drug: Placebos — Isotonic saline
  Arms: Placebo; Treatment B:

SUMMARY:
Dexamethasone twice for pain treatment after total knee arthroplasty - A Placebo-controlled, randomised, parallel 3-group multicentre trial of one and two doses of dexamethasone for postoperative treatment

DETAILED DESCRIPTION:
Trial name: Dexamethasone twice for pain treatment of total knee arthroplasty - A randomized blinded placebo-controlled clinical trial

Trial Acronym: DEX-2-TKA

Background: Effective postoperative pain management is essential for the well-being and rehabilitation of the surgical patient. No "gold standard" exists for pain treatment after total knee arthroplasty (TKA) since combinations of different analgesic treatments are used with nearly no evidence for combined analgesic efficacy. A single perioperative dose of glucocorticoid (GCC) (i.e. dexamethasone) has well established effects on postoperative nausea and vomiting, and may be beneficial for postoperative pain. A recent trial suggested that an additional postoperative dose of GCC improved postoperative pain treatment. Recent systematic reviews, sub-studies of RCTs and cohort studies of perioperative GCC raised no concern regarding serious adverse events of a single dose GCC for non-cardiac surgery. However, optimal dose, combination and regimen of perioperative GCC remains unsettled.

Objective: To establish the analgesic effect and safety of one and two consecutive days of a single dose of dexamethasone after TKA. GCC will be administered in combination with paracetamol, NSAID (ibuprofen), and local infiltration analgesia.

Intervention: The participants will be randomised in three groups: A) 24 mg dexamethasone i.v. perioperative (POD0) and 24 mg dexamethasone i.v. on the first postoperative day (POD1); B) 24 mg dexamethasone i.v. POD0 and placebo (isotonic saline) i.v. on POD1; and C) placebo i.v. on POD0 and POD1.

Design and trial size: Placebo-controlled, randomised, parallel 3-group multicentre trial with adequate centralised computer-generated allocation sequence and allocation concealment with unknown block size. Assessor, investigator, caregivers and participants will all be blinded. A total of 423 eligible participants are needed to detect a difference of 10 mg morphine for the first 48 hours postoperatively with a standard deviation of 23 mg, an overall familywise type 1 error rate of 0.05 and a type 2 error rate of 0.10. To compensate for uncertainty of the distribution a surplus of 15 % is added, thus a total of 486 patients will be included. To maintain an overall familywise error rate of 0.05 the sample size estimation is based on pairwise comparisons of the primary outcome between the three groups (three comparisons) with an individual type I error rate of 0.0167.

Sub studies: The investigators plan the following substudies

* One-year follow-up with EQ-5D-5L (EuroQuols - 5 dimension - 5 level score), Oxford-Knee-Score and mortality including need for medical attention.
* Troponin (TnI) levels 24 and 48 hours postoperatively (only at Naestved Hospital).
* Analysis of high and low pain responders.
* Establishment of a bio-bank (blood-samples) for future studies (only at Naestved Hospital).

Due to decisions made by the Steering Committee at our meeting the 14th of May 2019 in Køge, Region Zealand, Denmark, the secondary outcomes have been rearranged and divided into secondary outcomes and other (eksplorative) outcomes. Furthermore an additional explorative endpoint is added: Number of patients with a permanent use of opioids 90 days after surgery.

No data was unblinded or analyzed to aid the decisions.

After the last patient was included, but prior to data analysis and unmasking, the Steering Committee decided to include the following explorative outcomes in the main article reporting results from this trial. The decision was made by consensus via email 4th of October 2020:

* proportion of participants with one or more severe adverse event (SAE), including death, within 90 days after surgery (SAE defined according to ICH-GCP-guidelines, except 'prolongation of hospitalisation')
* opioid related adverse events (AE)

  * level of nausea, sedation and dizziness at 24 and 48 h
  * number of vomiting episodes 0-24 and 24-48 h"
  * use of anti-emetics 0-24 and 24-48 h

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral, primary total knee arthroplasty
* ASA 1-3
* BMI ≥ 18.0 and ≤ 40.0
* Negative urine HCG pregnancy test and use of anti-conception for women in the fertile age
* Patients who gave their written informed consent to participating in the trial after having fully understood the contents of the protocol and restrictions

Exclusion Criteria:

* Patients who cannot cooperate with the trial
* Concomitant participation in another trial involving medication
* Patients who cannot understand or speak Danish
* Patients with allergy to medication used in the trial
* Patients with daily use of high dose opioid (> oral morphine 30 mg/day or oxycodone 30 mg/day or tramadol 150 mg/day) or any use of other opioids including methadone and transdermal opioids.
* Patients with at daily use of systemic glucocorticoids
* Contraindications against ibuprofen or paracetamol, for example previous ulcer, known heart failure, known liver failure, or known renal failure (eGRF < 60 ml/kg/1,73m2), known thrombocytopenia (<100 bil/l); or against treatment with glucocorticoids.
* Dysregulated diabetes (investigators judgement)
* Patients suffering from alcohol and/or drug abuse - based on the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Cumulative usage of morphine 0-48 hours postoperatively | 0-48 hours postoperatively
  Morphine administered both as patient-controlled analgesia (PCA) i.v. morphine 0-24 hours and oral morphine on demand 24-48 hours, and any other supplemental morphine administered postoperatively.
  Consumption in mg

SECONDARY OUTCOMES:
VAS-pain scores (visual analogue scale (VAS)) | 24 and 48 hours postoperatively
  * with active 45 degrees flexion of the knee (VAS) at 24 and 48 hours postoperatively
  * at rest at 24 and 48 hours postoperatively
  * highest score during 0-24 hours and 24-48 hours
Adverse events, patient-reported | 0-48 hours postoperatively
  Number of patients with one or more patient-reported adverse event in the intervention period

OTHER OUTCOMES:
Number of patients with one or more serious adverse events (SAE) | 90 days postoperatively
  Number of patients with one or more serious adverse events (SAE), including death, within 90 days after surgery defined as SAE (according to ICH-GCP-guidelines), except "prolongation of hospitalisation"
90 days follow-up | 90 days postoperatively
  Number of patients with need for medical attention and/or intervention including need for anti-biotics and/or re-operation
Total need of i.v. morphine 0-24 hours postoperatively | 0-24 hours postoperatively
  Consumption in mg
Total need of oral morphine 24-48 hours postoperatively | 24-48 hours postoperatively
  Consumption in mg
VAS-pain scores (visual analogue scale (VAS)) | 6, 24 and 48 hours postoperatively hours postoperatively
  * with active 45 degrees flexion of the knee (VAS) at 6 hours postoperatively
  * at rest at 6 postoperatively
  * average score during 0-24 hours and 24-48 hours
Timed up and go (TUG) test at 24 and 48 hours including maximum pain during the TUG test. | 24 and 48 hours postoperatively
  The timed up and go test is performed at 24 and 48 hours postoperatively. The participant will be placed on a chair, 3 meters from a line. After the command "Go" the participant will
  1. Stand up from the chair
  2. Walk to the line on the floor
  3. Turn
  4. Walk back to the chair
  5. Sit down again.
  The time will be measured from "Go" to the participant is sitting again.
Adverse events, nausea | 0-48 hours postoperatively
  Level of nausea at 6, 24 and 48 hours postoperatively
  Scale: none, mild, moderate, severe
Adverse events, sedation | 0-48 hours postoperatively
  Level of sedation at 6, 24 and 48 hours postoperatively
  Scale: none, mild, moderate, severe
Adverse events, dizziness | 0-48 hours postoperatively
  Level of dizziness at 6, 24 and 48 hours postoperatively
  Scale: none, mild, moderate, severe
Adverse events, vomiting | 0-48 hours postoperatively
  Number of vomiting episodes (0-48 hours) measured in the periods 0-24 and 24-48 hours postoperatively
Consumption of antiemetics in the period 0-24 and 24-48 hours postoperatively | 0-48 hours postoperatively
  Use of ondansetron and DHB (Dehydrobenzperidol)
Quality of sleep 0-24 and 24-48 hours postoperatively | 0-48 hours postoperatively
  Scale: very bad, fairly bad, fairly good, very good
Level of fatigue at 24 and 48 hours postoperatively | 24 and 48 hours postoperatively
  Scale: none, mild, moderate, severe
NRS-pain scores 3-7 days postoperatively | 3-7 days postoperatively
  Two daily NRS-scores: One in the morning and one in the evening
Quality of sleep 3-7 days postoperatively | 3-7 days postoperatively
  Scale: very bad, fairly bad, fairly good, very good
Satisfaction with postoperative pain treatment after 7 days | 7 days postoperatively
  Scale: very bad, fairly bad, fairly good, very good
Proportion of participants with permanent use of opioids 90 days after surgery | 90 days postoperatively
  Number of patients with prescripción for painkillers
90 days follow-up using EQ5D5L | 90 days postoperatively
  Qualitative participant reported assessments using EQ5D5L (Questionaire - with one NRS (0-100))
90 days follow-up using Oxford-Knee-Score | 90 days postoperatively
  Qualitative participant reported assessments using Oxford-Knee-Score (Questionaire, scale 12-60 points)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, PhD, Assoc Prof, Study Chair — Department of Anaesthesiology, Zealand University Hospital, Køge; Daniel Hägi-Pedersen, MD, PhD, Study Chair — Department of Anaesthesiology, Næstved Hospital; Jørgen B Dahl, DMSc, Study Chair — Department of Anaesthesiology, Bispebjerg Hospital; Kasper S Gasbjerg, MD, Principal Investigator — Department of Anaesthesiology, Næstved Hospital; Troels H Lunn, DMSc, Study Chair — Department of Anaesthesiology, Bispebjerg Hospital
Locations (5):
- Denmark (5):
  - Gildhøj Privathospital, Brøndby
  - Bispebjerg Hospital, Copenhagen
  - Sjællands Universitetshospital, Køge, Køge
  - Næstsved Sygehus, Næstved
  - Odense Universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Data will also be published anonymised according to ICIMEs (International Committee of Medical Journal Editors) guidelines
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Molgaard AK, Gasbjerg KS, Mathiesen O, Hagi-Pedersen D, Gogenur I. Dexamethasone vs. placebo modulation of the perioperative blood immune proteome in patients undergoing total knee arthroplasty. BMC Anesthesiol. 2025 Mar 21;25(1):136. doi: 10.1186/s12871-025-03003-3. PMID 40119286
- [Derived] Derby CB, Gasbjerg KS, Hagi-Pedersen D, Lunn TH, Pedersen NA, Lindholm P, Brorson S, Schroder HM, Thybo KH, Bagger J, Lindberg-Larsen M, Overgaard S, Jakobsen JC, Mathiesen O. Prolonged effects of dexamethasone following total knee arthroplasty: A pre-planned sub-study of the DEX-2-TKA trial. Acta Anaesthesiol Scand. 2024 Jan;68(1):35-42. doi: 10.1111/aas.14319. Epub 2023 Sep 14. PMID 37709280
- [Derived] Gasbjerg KS, Hagi-Pedersen D, Lunn TH, Laursen CC, Holmqvist M, Vinstrup LO, Ammitzboell M, Jakobsen K, Jensen MS, Pallesen MJ, Bagger J, Lindholm P, Pedersen NA, Schroder HM, Lindberg-Larsen M, Norskov AK, Thybo KH, Brorson S, Overgaard S, Jakobsen JC, Mathiesen O. Effect of dexamethasone as an analgesic adjuvant to multimodal pain treatment after total knee arthroplasty: randomised clinical trial. BMJ. 2022 Jan 4;376:e067325. doi: 10.1136/bmj-2021-067325. PMID 34983775
- [Derived] Gasbjerg KS, Hagi-Pedersen D, Lunn TH, Overgaard S, Pedersen NA, Bagger J, Lindholm P, Brorson S, Schroder HM, Thybo KH, Mathiesen O, Jakobsen JC. DEX-2-TKA - DEXamethasone twice for pain treatment after Total Knee Arthroplasty: Detailed statistical analysis plan for a randomized, blinded, three-group multicentre clinical trial. Acta Anaesthesiol Scand. 2020 Jul;64(6):839-846. doi: 10.1111/aas.13560. Epub 2020 Mar 3. PMID 32048274
- [Derived] Gasbjerg KS, Hagi-Pedersen D, Lunn TH, Jakobsen JC, Overgaard S, Pedersen NA, Bagger J, Lindholm P, Brorson S, Schroder HM, Thybo KH, Mathiesen O. DEX-2-TKA-DEXamethasone twice for pain treatment after Total Knee Arthroplasty: A protocol for a randomized, blinded, three-group multicentre clinical trial. Acta Anaesthesiol Scand. 2020 Feb;64(2):267-275. doi: 10.1111/aas.13481. Epub 2019 Oct 18. PMID 31544230